CLINICAL TRIAL: NCT02868762
Title: Correlation of the Neck Disability Index (NDI) and Voice Handicap Index (VHI) in Neck Pain Patients and Patients With Voice Disorders
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BJ_23_03_2016
Record Dates: First submitted 2016-07-04; First posted 2016-08-16 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Neck Pain and/or a Voice Disorder
Keywords: neck pain, voice disorder
MeSH Terms: conditions — Neck Pain; Voice Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This study investigates in patients whose primary complaint is either neck pain and/or a voice disorder , if there are any correlations between subjective neck and voice symptoms according to Neck Disability Index (NDI) and Voice Handicap Index (VHI). NDI and VHI questionnaire results for voice disordered patients will be retrieved from the data base of the Department of Phoniatrics and Speech Pathology, University Hospital Zurich. Neck pain patient questionnaire data will be retrieved from an ongoing study. The agreement between subjective neck handicap (NDI) and voice handicap (VHI) will be statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* primary diagnose of a functional disorder of the muscular structure in the neck area
* primary diagnose of a functional or secondary structural voice disorder

Exclusion Criteria:

* systemic illness of the motion apparatus (i.e., polyarthritis rheumatica)
* acute cancer
* neurogenic voice and swallow disorder
* Intubation within the last 18 months
* lack of german knowledge, (not able to fill out a questionnaire independently)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic patients
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Correlation between neck disability index and voice handicap index (questionnaire) | 1 day

SECONDARY OUTCOMES:
Additional neck area handicap in patients with voice disorders (questionnaire) | 1 day
  Patients will fill out the questionnaire once, at the beginning of the study
Additional subjective voice disorder in patients with neck pain (questionnaire) | 1 day
  Patients will fill out the questionnaire once, at the beginning of the study
Difference in pain strength and quality in patients with functional voice disorder as compared to patients with benign organical vocal fold changes (questionnaire) | 1 day
  Patients will fill out the questionnaire once, at the beginning of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Bohlender, KD Dr., Principal Investigator — University Hospital Zurich, clinic othorhinolaryngology, 8091 Zurich
Locations (1):
- KD Dr. Jörg Bohlender, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No